CLINICAL TRIAL: NCT03653689
Title: Molecular Phenotyping of IBS Subtypes
Brief Title: Identification of IBS Metabotypes Based on Physiological Responses to Food
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Chalmers University of Technology (Other)
Responsible Party: Principal Investigator, Per Hellström, Medical doctor, Professor, Uppsala University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: OpDiMet1
Record Dates: First submitted 2018-08-19; First posted 2018-08-31 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; metabotype; FODMAP; gluten
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet; Glutens

STUDY DESIGN:
Intervention Model Description: The study will be a double-blinded, randomized, placebo-controlled cross-over study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study will be double-blinded. Neither the participant nor the care providers or the outcome assessor will know which treatment is which.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FODMAPs (Active Comparator): Dietary supplement: FODMAPs 50 grams three servings per day for seven days.
  Interventions: Dietary Supplement: FODMAP; Dietary Supplement: Gluten; Dietary Supplement: Placebo
- Gluten (Active Comparator): Dietary supplement: Gluten 17.3 grams three servings per day for seven days.
  Interventions: Dietary Supplement: FODMAP; Dietary Supplement: Gluten; Dietary Supplement: Placebo
- Placebo (Placebo Comparator): Dietary supplement: Placebo rice porrige three servings per day for seven days.
  Interventions: Dietary Supplement: FODMAP; Dietary Supplement: Gluten; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: FODMAP — The intervention will run for seven weeks. During the whole intervention, the participants will hold a baseline diet with no gluten and low intake of FODMAPs. The first week, the participants will consume a one-time cocktail provocation consisting of gluten (17.3 gram) and FODMAPs (50 gram) Thereafter, study participants will receive three 1-week diets with additions of either FODMAPs, gluten or an inert control with 1-week washout in-between. The daily amount for gluten will be 17.3 gram and the daily amount for FODMAPs will be 50 gram. The order of the three weeks with extra diets (gluten/FODMAPs/control) will be randomized.
Dietary Supplement: Gluten — The intervention will run for seven weeks. During the whole intervention, the participants will hold a baseline diet with no gluten and low intake of FODMAPs. The first week, the participants will consume a one-time cocktail provocation consisting of gluten (17.3 gram) and FODMAPs (50 gram) Thereafter, study participants will receive three 1-week diets with additions of either FODMAPs, gluten or an inert control with 1-week washout in-between. The daily amount for gluten will be 17.3 gram and the daily amount for FODMAPs will be 50 gram. The order of the three weeks with extra diets (gluten/FODMAPs/control) will be randomized.
Dietary Supplement: Placebo — The intervention will run for seven weeks. During the whole intervention, the participants will hold a baseline diet with no gluten and low intake of FODMAPs. The first week, the participants will consume a one-time cocktail provocation consisting of gluten (17.3 gram) and FODMAPs (50 gram) Thereafter, study participants will receive three 1-week diets with additions of either FODMAPs, gluten or an inert control with 1-week washout in-between. The daily amount for gluten will be 17.3 gram and the daily amount for FODMAPs will be 50 gram. The order of the three weeks with extra diets (gluten/FODMAPs/control) will be randomized.

SUMMARY:
Irritable bowel syndrome (IBS) is a condition characterized by abdominal pain, bloating, constipation, diarrhea and gas and affects up to 15% of the Western population. In many individuals with IBS, symptoms can be triggered by foods, such as FODMAPs (easily fermentable dietary fiber containing Fermentable Oligosaccharides, Disaccharides, Monosaccharides, and Polyols). Some individuals with IBS may also benefit from a gluten-free diet. Current subtypes of IBS are based on symptoms (constipation, diarrhea, and mixed), rather than mechanistic differences. Another promising approach for identifying IBS subtypes is based on grouping individuals into similar metabolic phenotypes, i.e. metabotypes, that share similarities in metabolism and metabolic regulation in response to specific foods. Health and wellbeing could potentially be improved by personalized treatment through tailoring diet to subjects with different IBS subtypes.

To investigate this hypothesis, the investigators will conduct an intervention study on subjects with IBS and identify specific food susceptibilities based on metabolic phenotype (metabotype). In total, 120 women and men with moderate to severe IBS will be recruited. Gluten intolerance, other gastrointestinal disease and abdominal surgery will constitute exclusion criteria. The study will be performed in a double-blind, randomized, placebo-controlled cross-over study design. Study participants will receive three 1-week diets with additions of either FODMAPs, gluten or an inert control with 1-week washout in-between. IBS metabotypes will be identified by integrative multivariate analysis of molecular phenotype data from metabolomics and microbiota measurements combined with data on bowel habits and stomach discomfort. Study participants will also be subjected to a cocktail provocation containing FODMAPs and gluten to develop a rapid diagnostic test based on identified plasma metabolomic biomarkers of IBS metabotypes.

DETAILED DESCRIPTION:
The current study is explorative with the primary aim to find and relate distinct subject metabotypes reflecting tolerance/intolerance to specific food components among IBS-patients by deducing and relating OMICs data patterns (metabolomics and gut microbiota data) to reported severity of IBS-symptoms indicated by the primary endpoint variable, i.e. IBS-SSS. Since the investigators don't have an estimation of the variation in the multivariate OMICs-data (both metabolomics and 16S rRNA analysis of bacterial RNA), it is not possible to perform an adequate power-calculation. There is a lack of consensus on how to best perform power analysis for these OMICs-designs (and therefore also a lack of tools), although some initiatives have been published. Power analysis is especially difficult in untargeted metabolomics, where the number of variables are not a priori determined, where there is strong multi-colinearity and where variables cannot be assumed to contribute with equal power to effect size. Moreover, there is a shortage of relevant untargeted metabolomics and microbiota study material on IBS x diet interactions from which to estimate relevant parameters such as multivariate effect sizes and variance estimates, due to the surprisingly few metabolomics studies on IBS and the total lack of publicly available raw data. However, significant differences in the metabolome was previously observed in children with or without diarrhea-dominant IBS (n=22 per group). Systematic differences were also shown in individual metabolites in persons with IBS consuming either a high or low FODMAP diet (n≈20 per treatment).

In this study, a cross-over design will be performed, which will increase the power compared to parallel designs. Moreover, participants will be stratified with respect to subtype of IBS (i.e. diarrhea, constipation and mixed). However, the investigators will not know in advance how many IBS-metabotypes will be present in the material or the quantitative distribution between the metabotypes. Therefore, 120 participants will be recruited to be able to observe significant differences between dietary treatments, based on the assumptions that it will be possible to identify around 4±1 metabotypes, and an approximate equal distribution between metabotypes (≥20 persons per metabotype). In addition, a selection of 120 participants will, under these conditions allow for 20% drop-out from the study, which is a high estimate based on our previous experience from nutritional interventions. An important secondary outcome from this study material is that it will give the opportunity to be used for power calculations in future OMICs-studies where the effect sizes on both clinical parameters and OMICs-measures are uncertain.

Discovery of IBS metabotypes Identification of metabotypes will be performed using predominantly multivariate data analytical techniques. During initial analyses, molecular phenotype data (metabolomics and microbiota) will be analyzed using unsupervised principal component analysis (PCA) and clustering techniques to investigate whether data self-aggregates into meaningful clusters. To adjust for between-individual variability and focus on the effects of interventions, variance partitioning (sometimes referred to as ANOVA decomposition) by individual will be performed. Clusters will be correlated with recorded IBS/clinical data (IBS-SSS, bowel emptying diary) to examine whether emerging clusters contain functional information in relation to IBS symptoms. Moreover, it is likely that different clusters are not similarly reflected in plasma and fecal metabolomics and fecal microbiota. To investigate to which extent the different clusters are associated with the different omics blocks, a series of techniques for subdivision of variability into common and distinct components will be applied to the unsupervised analysis.

In a second line of unsupervised analysis, PCA and clustering analyses will be performed on molecular phenotype aggregated with IBS/clinical data, which will have the potential to influence clustering directly instead of investigating correlations afterwards. Again, subdivision of variability into common and distinct components will be applied to examine how clusters are reflected in the different data blocks.

Finally, supervised analyses will be used to directly associate molecular phenotype data (independent variables) with IBS/clinical data (dependent variables) using in-house developed partial least squares (PLS) and random forest (RF) techniques. These in-house techniques are specifically adapted to identifying the most relevant set of independent variables to describe the covariability with the dependent data (submitted manuscript). IBS/clinical data can be used both as continuous multiple variables or directly by converting observations to clusters. To examine how clusters and IBS/clinical data are reflected in the different omics blocks, newly developed procedures to find common and distinct components in supervised analysis will be applied (submitted manuscript).

The progression in these three approaches represent an increasing degree of supervision in multivariate analysis. After all analyses, emerging clusters from the PCA and clustering analyses and multivariate predictions from the PLS and RF analyses will further analyzed using bioinformatics tools adapted to provide meaningful biological interpretation with the aim to confirm correspondence between clusters and metabotypes.

Rapid diagnostic test of metabotypes After metabotypes have been identified, multivariate predictive analysis of the mixed gluten/FODMAP exposure will be performed to identify predictive biomarkers of metabotypes. These models will similarly as above be based on in-house PLS and RF procedures using metabolomics data as independent variables and metabotype classification per individual as dependent variable.

Plasma metabolic profiles will be analyzed regularly up to 4 hours post exposure and two different approaches will be undertaken to address the time-trends in metabolic profiling: In a first approach, time profiles will be converted to areas-under-the-curve per measured metabolite feature through numerical integration. These values will then be used directly as independent variables to give an indication of overall reflection of metabotype on metabolite levels after exposure. However, this direct approach will not be able to take into consideration potential differences in time-trends between metabotypes. Therefore, variance partitioning hyphenated with supervised learning will be used to investigate metabotype x time interactions. This approach will require method development in multivariate analysis, which is currently underway in the R Landbergs research group and expected to be ready and beta-tested during 2018, i.e. before data is available for analysis. This methodology is projected to allow for simultaneous analysis of overall differences in metabolite levels between treatments as well as differences in time profiles, thereby giving information also on the most opportune time points to draw samples for effective prediction of metabotype x.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Men and women
* Medium to severe IBS
* Age 18-70 years
* BMI 18.5-38 kg/m2
* Hb 120-160 g/L
* S-TSH <4 mIU/L
* S-CRP <5 mg/L
* S-Transglutaminase IgA <7 U/mL
* Willingness to consume rice porridge, once a day for 3 weeks
* Any medication stable for the last 14 days.

Exclusion Criteria:

* Gluten intolerance
* Other gastrointestinal disease (e.g. Crohn's disease, ulcerative colitis)
* Performed bariatric surgery
* Previous abdominal surgery, other than appendectomy.
* Food adaptation (eg. vegetarian, LCHF) in order to achieve abdominal relief
* Medical treatment for weight reduction.
* ≥10 kg of weight change in the last 12 months
* Diastolic blood pressure more than 105 mm Hg at visit 1
* Systolic blood pressure more than 160 mm at visit 1
* Blood donation or participation in a clinical study with blood sampling within 30 days prior to screening visit and throughout the study
* Pregnant or lactating or wishes to become pregnant during the period of the study.
* Pharmacological medication with drugs known to possibly affect gastrointestinal function, eg antidepressants, neuroleptics, proton pump inhibitors, H2-receptor blockers, non-steroidal anti-inflammatory drugs, opioids, loperamide, cholestyramine, laxatives, metoclopramide, domperidone, prucalopride, linaclotide
* Unstable pharmacological medication
* History of drug or alcohol abuse
* Using nicotine products on a daily basis (incl. chewing gum, patches, snus etc.)
* Lack of suitability for participation in the trial, for any reason, as judged by the medical doctor or PI.
* Unable to understand written and spoken Swedish language.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
IBS-SSS | When the study is completed, anticipated in 1-2 year
  The questionnaire IBS-SSS will be used to monitor the IBS symptoms and relate it to how participants metabolically react to the diets (gluten, FODMAPS and control). The IBS-SSS will also be related to how the microbiota potentially could differentiate between individuals and how it can be related to the diets (gluten, FODMAPS and control).

SECONDARY OUTCOMES:
BMI | When the study is completed, anticipated in 1-2 year
  Body weight (kg) and height (meters) will be combined to report BMI in kg/m^2. It will be related to IBS subtypes and how participants react on the diets (gluten, FODMAPS and control)
Blood pressure | When the study is completed, anticipated in 1-2 year
  Blood pressure (mmHg) will be related to the IBS subtypes and how participants react on the diets (gluten, FODMAPS and control)
Heart rate | When the study is completed, anticipated in 1-2 year
  Heart rate (bpm) will be related to the IBS subtypes and how participants react on the diets (gluten, FODMAPS and control)

CONTACTS AND LOCATIONS:
Overall Officials: Per Hellström, Prof, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data will be available after data base lock.
Time Frame: After September 2020.
Access Criteria: Data sharing for supplement data on publication.

REFERENCES:
- [Result] Shankar V, Reo NV, Paliy O. Simultaneous fecal microbial and metabolite profiling enables accurate classification of pediatric irritable bowel syndrome. Microbiome. 2015 Dec 9;3:73. doi: 10.1186/s40168-015-0139-9. PMID 26653757
- [Result] McIntosh K, Reed DE, Schneider T, Dang F, Keshteli AH, De Palma G, Madsen K, Bercik P, Vanner S. FODMAPs alter symptoms and the metabolome of patients with IBS: a randomised controlled trial. Gut. 2017 Jul;66(7):1241-1251. doi: 10.1136/gutjnl-2015-311339. Epub 2016 Mar 14. PMID 26976734
- [Derived] Nordin E, Landberg R, Hellstrom PM, Brunius C. Exploration of differential responses to FODMAPs and gluten in people with irritable bowel syndrome- a double-blind randomized cross-over challenge study. Metabolomics. 2024 Feb 12;20(2):21. doi: 10.1007/s11306-023-02083-x. PMID 38347192
- [Derived] Nordin E, Hellstrom PM, Vuong E, Ribbenstedt A, Brunius C, Landberg R. IBS randomized study: FODMAPs alter bile acids, phenolic- and tryptophan metabolites, while gluten modifies lipids. Am J Physiol Regul Integr Comp Physiol. 2023 Sep 1;325(3):R248-R259. doi: 10.1152/ajpregu.00016.2023. Epub 2023 Jul 3. PMID 37399002
- [Derived] Nordin E, Hellstrom PM, Brunius C, Landberg R. Modest Conformity Between Self-Reporting of Bristol Stool Form and Fecal Consistency Measured by Stool Water Content in Irritable Bowel Syndrome and a FODMAP and Gluten Trial. Am J Gastroenterol. 2022 Oct 1;117(10):1668-1674. doi: 10.14309/ajg.0000000000001942. Epub 2022 Aug 12. PMID 36087104
- [Derived] Nordin E, Brunius C, Landberg R, Hellstrom PM. Fermentable oligo-, di-, monosaccharides, and polyols (FODMAPs), but not gluten, elicit modest symptoms of irritable bowel syndrome: a double-blind, placebo-controlled, randomized three-way crossover trial. Am J Clin Nutr. 2022 Feb 9;115(2):344-352. doi: 10.1093/ajcn/nqab337. PMID 34617561